CLINICAL TRIAL: NCT01109472
Title: Improving Osteoporosis Care in a Home Health Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eli Lilly and Company (Industry); Alacare Home Health and Hospice (Other)
Responsible Party: Principal Investigator, Jeff Curtis, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: X080401004; B3D-US-X016 (Other Grant/Funding Number: Eli Lilly and Company)
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient Tailored Magazine (Experimental): Patient responses from computer assisted telephone interviews will be used to develop a patient tailored educational magazine.
  Interventions: Other: patient magazine

INTERVENTIONS:
Other: patient magazine — patient magazine individually tailored to patient's prior feedback

SUMMARY:
Study aims to improve osteoporosis care through patient tailored education materials in a group-randomized trial of patients referred to home health care with a history of fracture and/or an osteoporosis diagnosis. Project investigators will conduct telephone surveys and examine electronic medical record data to assess fracture related morbidity and mortality, osteoporosis treatment and adherence, and use of calcium and vitamin D supplements.

We hypothesize that patients that receive the intervention materials will be more likely to initiate or maintain osteoporosis treatment.

ELIGIBILITY:
Inclusion Criteria:

* prior fracture
* osteoporosis diagnosis
* received home health care

Exclusion Criteria:

* hospice
* active cancer treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1009 (Actual)
Dates: Start 2009-04; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Initiation/Maintenance of Anti-osteoporosis prescription medication | Three months post initial survey

SECONDARY OUTCOMES:
Initiation/Maintenance of calcium and vitamin D | Three months post initial survey

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Curtis, MD, MPH, Principal Investigator — University of Alabama at Birmingham